CLINICAL TRIAL: NCT03064568
Title: Rectal Misoprostol as a Hemostatic Agent During Abdominal Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC20150554H
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myomectomy; Surgical Blood Loss
Keywords: Myomectomy, Misoprostol, Vasopressin, Blood loss
MeSH Terms: conditions — Blood Loss, Surgical; Diabetes Insipidus; Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Prospective double-blinded study completed at a tertiary care center
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization to treatment arm done by 3rd party. Randomization will be performed by a third party so that neither the surgeon nor patient will know which intervention was performed, and interventions will be placed in sealed, sequentially numbered, opaque envelopes. The code will only be broken at time of data analysis once all patients have been enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Misoprostol 200Mcg Tab (Experimental): Patients will receive misoprostol 800mcg per rectum 30 minutes preoperatively.
  Interventions: Drug: Misoprostol 200Mcg Tab
- Placebo (Placebo Comparator): Patients will receive identical inert tablets per rectum 30 minutes preoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol 200Mcg Tab — 4 tablets will be inserted rectally
  Other Names: Cytotec
  Arms: Misoprostol 200Mcg Tab
Drug: Placebo
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
Purpose is to identify if misoprostol in addition to local vasopressin decreases blood loss when compared to vasopressin alone, which is our current practice at this time. The study will be double-blinded with neither the patient nor the researcher knowing whether the placebo or the misoprostol was given. We will monitor patients for decrease in hemoglobin and hematocrit, need for transfusion, and operative time among other measures of perioperative morbidity to see if the addition of misoprostol makes a significant difference. We will also observe patients to see if there are any side effects of misoprostol that make its use undesirable.

DETAILED DESCRIPTION:
All women with planned myomectomy receive Depo Leupron prior to surgery per standard care and undergo routine pre-operative laboratory testing including hemoglobin and hematocrit. If enrolled in the study, patients will be consented at their pre-op appointment for the study and be asked to complete a visual analog scale to assess pre-operative pain. Patients will be randomized to receive misoprostol 800mcg per rectum or an identical inert tablet(s) per rectum 30 minutes preoperatively. Randomization will be performed by a third party so that neither the surgeon nor patient will know which intervention was performed, and interventions will be placed in sealed, sequentially numbered, opaque envelopes. Researcher team will have all needed data corresponding with randomized code which will be broken at conclusion of study and will be able to match code with patient's initials and medical record number after study completion to analyze data. Myomectomy will then be performed per standard care with the use of local vasopressin to aid in decreasing blood loss per our normal standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Female age 20-50 y/o who plan to undergo abdominal myomectomy for symptomatic myomatous uterus

Exclusion Criteria:

* Patient with contraindication to misoprostol or vasopressin, personal history or cardiac or pulmonary disease, history of prior myomectomy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patient must have a uterus to participate
Enrollment: 18 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randal M Robinson, MD, Principal Investigator — UT Health San Antonio
Locations (3):
- United States (3):
  - St. Lukes Baptist Hospital, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no significant pre-assignment procedures beyond standard preoperative care and consent. Before randomization, patients undergo a physical exam, transvaginal ultrasound, receive Depo Leupron, have preoperative hemoglobin and hematocrit testing, and complete a preoperative pain assessment after providing consent.
Groups:
- Misoprostol 200Mcg Tab: Patients will receive misoprostol 800mcg per rectum 30 minutes preoperatively.
  Misoprostol 200Mcg Tab x4
- Placebo: Patients will receive identical inert tablets per rectum 30 minutes preoperatively.
  Placebo
Period: Overall Study
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who receive an abdominal myomectomy
Groups:
- Misoprostol 200Mcg Tab: Patients will receive misoprostol 800mcg per rectum 30 minutes preoperatively.
  Four Misoprostol 200Mcg Tab
- Total: Total of all reporting groups
Arm/Group | Misoprostol 200Mcg Tab | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Customized [Count of Participants; unit: Participants]
  20-50 years of age | 8 | 10 | 18
Sex/Gender, Customized [Count of Participants; unit: Participants] — All participants were female
  Participants
    Female | 8 | 10 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Surgical Blood Loss
Description: Estimated blood loss during surgery
Time Frame: Intraoperative
Population: Participants who receive an abdominal myomectomy
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Number analyzed (Participants) | 8 | 10
ml | 761 (504) | 691 (532)

2. Secondary Outcome: Febrile Morbiditiy
Description: Number of participants that have evidence of fever or infection postoperatively
Time Frame: 24 hours postop
Population: Participants who receive an abdominal myomectomy
Measure: Number; unit: participants
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Number analyzed (Participants) | 8 | 10
participants | 0 | 0

3. Secondary Outcome: Need for Blood Transfusion
Description: Number of participants that had a requirement of blood transfusion
Time Frame: intraoperative to 24 hours postoperative
Population: Participants who receive an abdominal myomectomy
Measure: Number; unit: participants
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Number analyzed (Participants) | 8 | 10
participants | 1 | 0

4. Secondary Outcome: Pain Score
Description: Assessment of patient subjective pain with the visual analog scale prior to discharge from hospital. The scale used is a a likert pain scale where the participant selects their pain level between 0- 10, where 10 is the highest level of pain experienced.
Time Frame: 24 hours postop
Population: Participants who receive an abdominal myomectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Number analyzed (Participants) | 8 | 10
score on a scale | 4.63 (2.39) | 4.65 (1.38)

5. Secondary Outcome: Number of Participants With Medication Side-effects
Description: Surveillance for any adverse side effects from misoprostol
Time Frame: 24 hours postop
Population: Participants who receive an abdominal myomectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 200Mcg Tab | Placebo
Number analyzed (Participants) | 8 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the immediate postoperative period, specifically within 24 hours after surgery and prior to hospital discharge.
Description: Postoperatively prior to discharge, patients were monitored in the hospital for 24 hours after surgery occured, up to 2 days total. During this period, hemoglobin and hematocrit were remeasured, pain was assessed, and patients were evaluated for side effects of misoprostol, including fever, chills, and diarrhea, prior to discharge.
Arm/Group | Misoprostol 200Mcg Tab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03064568/Prot_SAP_000.pdf